CLINICAL TRIAL: NCT01299688
Title: HER2 Circulating Tumor Cells in Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Professor, Samsung Medical Center
Other Study IDs: 2009-12-008
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, circulating tumor cell
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to survey the frequency of HER2 (+) CTC in order to lay groundwork for future clinical trials incorporating Her-2 targeted agents in gastric cancer.

DETAILED DESCRIPTION:
We propose to survey the frequency of HER2 (+) CTC in order to lay groundwork for future clinical trials incorporating Her-2 targeted agents in gastric cancer. Blood samples will be collected from metastatic gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years ② Patients with localized, histologically confirmed gastric cancer ③ Informed consent form

Exclusion Criteria:

* No informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2013-03-11 (Actual); Study Completion 2013-03-11 (Actual)

PRIMARY OUTCOMES:
To survey the frequency of HER2(+) CTC in gastric cancer | 24month

CONTACTS AND LOCATIONS:
Overall Officials: Won Ki Kang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea